CLINICAL TRIAL: NCT06564987
Title: Risk of Nerve Damage After Administration of an Inferior Alveolar Nerve Block Using 4% Articaine Versus 2% Lidocaine
Brief Title: Risk of Nerve Damage After Administration of Local Anesthesia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDIOS0005
Record Dates: First submitted 2024-07-26; First posted 2024-08-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Inferior Alveolar Nerve Injuries
MeSH Terms: conditions — Mandibular Nerve Injuries | interventions — Carticaine; Epinephrine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Articaine (Experimental): Inferior Alveolar Nerve block using Articaine 4% with 1:200,000 epinephrine local anesthetic
  Interventions: Drug: 4% Articaine with 1:200,000 epinephrine
- Lidocaine (Active Comparator): Inferior Alveolar Nerve block using 2% lidocaine with 1:100,000 epinephrine local anesthetic
  Interventions: Drug: 2% lidocaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 4% Articaine with 1:200,000 epinephrine — Inferior Alveolar Nerve Block with 4% articaine
  Arms: Articaine
Drug: 2% lidocaine with 1:100,000 epinephrine — Inferior Alveolar Nerve Block with 2% lidocaine
  Arms: Lidocaine

SUMMARY:
This research aims to evaluate of the risk of nerve damage following the administration of articaine 4% and lidocaine 2% for Inferior Alveolar nerve Block (IANB). A Randomized Controlled Clinical Trial will be conducted where the patient will be randomly assigned to one the two groups; articaine 4% and Lidocaine 2%. The type of LA will be concealed to the operator, investigators and assessors. The patients will be monitored for any aigns of nerve parathesia for 3 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18-55 years old
* Patients need IANB
* healthy patient

Exclusion Criteria:

* medical conditions
* allergies
* medications
* pregnancy and breastfeeding
* inability to provide informed consent
* specific dental or medical history.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Electromyograph | 3 months
  Signs of loss of sensation in the involved side of the jaw will be recorded using a tool called Electromyograph machine to evaluate and record Nerve conduction velocity, the scale is as follow Normal (grade 0) to extremely damage of (grade 6) while a patient rate pain intensity on a Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Hashem, PhD, Study Director — Cleveland Dental Institute; Waleed Elmallah, PhD, Principal Investigator — Cleveland Dental Institute
Locations (2):
- United States (2):
  - Cleveland Dental Institute, Akron, Ohio
  - Cleveland Dental Institute, Ashtabula, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pogrel MA, Thamby S. Permanent nerve involvement resulting from inferior alveolar nerve blocks. J Am Dent Assoc. 2000 Jul;131(7):901-7. doi: 10.14219/jada.archive.2000.0308. PMID 10916328
- [Result] Mikesell P, Nusstein J, Reader A, Beck M, Weaver J. A comparison of articaine and lidocaine for inferior alveolar nerve blocks. J Endod. 2005 Apr;31(4):265-70. doi: 10.1097/01.don.0000140576.36513.cb. PMID 15793381
- [Result] Katyal V. The efficacy and safety of articaine versus lignocaine in dental treatments: a meta-analysis. J Dent. 2010 Apr;38(4):307-17. doi: 10.1016/j.jdent.2009.12.003. Epub 2009 Dec 16. PMID 20006669
- [Result] Stirrup P, Crean S. Does articaine, rather than lidocaine, increase the risk of nerve damage when administered for inferior alveolar nerve blocks in patients undergoing local anaesthesia for dental treatment? A mini systematic review of the literature. Br Dent J. 2019 Feb 8;226(3):213-223. doi: 10.1038/sj.bdj.2019.98. PMID 30734772
- [Result] Hook H. Inferior alveolar nerve block: is articaine better than lidocaine? Br Dent J. 2021 May;230(9):579-582. doi: 10.1038/s41415-021-2941-z. Epub 2021 May 14. PMID 33990740
- [Result] Samdrup T, Kijsamanmith K, Vongsavan K, Rirattanapong P, Vongsavan N. The effect of inferior alveolar nerve block anesthesia of 4% articaine and epinephrine 1:100,000 on blood flow and anesthesia of human mandibular teeth. J Dent Sci. 2021 Jan;16(1):249-255. doi: 10.1016/j.jds.2020.05.013. Epub 2020 Jun 4. PMID 33384805
- [Result] Aquilanti L, Mascitti M, Togni L, Contaldo M, Rappelli G, Santarelli A. A Systematic Review on Nerve-Related Adverse Effects following Mandibular Nerve Block Anesthesia. Int J Environ Res Public Health. 2022 Jan 31;19(3):1627. doi: 10.3390/ijerph19031627. PMID 35162650